CLINICAL TRIAL: NCT04722432
Title: Evaluation of Deployment Capability and Accuracy of an Outside the Scope (OTS), Detachable Catheter System for Ablation of Peripheral Lung Lesions: An Ex-Vivo Human Lung Model Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre hospitalier de l'Université de Montréal (CHUM) (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CE 20.220
Record Dates: First submitted 2020-10-16; First posted 2021-01-25 (Actual); Last update posted 2024-02-02 (Actual); Status verified 2024-02

CONDITIONS: Lung Cancer
MeSH Terms: conditions — Lung Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Système de cathéter détachable dehors du scope (DDS) (Experimental)
  Interventions: Device: Outside the Scope (OTS), Detachable Catheter System

INTERVENTIONS:
Device: Outside the Scope (OTS), Detachable Catheter System — Evaluation of Deployment Capability and Accuracy of an Outside the Scope (OTS), Detachable Catheter System for Ablation of Peripheral Lung Lesions: An Ex-Vivo Human Lung Model Study

SUMMARY:
A novel OTS detachable probe system carried outside and along the flexible bronchoscope has been developed. Using this novel system, the operator can deploy the probe in the target bronchus and lesion and completely detach the scope from the probe.

DETAILED DESCRIPTION:
Lung ablative therapies have growing interest in the treatment of early-stage primary lung cancer in surgical high-risk patients and as part of multimodal treatment in patients with large lesions or metastatic malignant disease in the lungs. Endobronchial ablative strategies allow deliver y of these therapies through a natural orifice and minimally invasive approach, potentially improving safety and reducing related morbidity. Application and deployment of this system allows the operator to have constant control of the airway, preventing life-threatening hemoptysis and other complications. We hypothesize that this novel detachable OTS system can be successfully deployed in the peripheral parenchymal target with potential clinical applications in the near future.

ELIGIBILITY:
Inclusion Criteria:

* Patients who follow surgery for the removal of diseased lungs before being submitted to a bilateral lung transplant.

Exclusion Criteria:

* None

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2020-10-16 (Actual); Primary Completion 2023-09-21 (Actual); Study Completion 2023-09-21 (Actual)

PRIMARY OUTCOMES:
accuracy of the deployment method | Time of procedure
  will be measured by bidimensional fluoroscopy images (antero-posterior and latero-lateral). The deployment will be considered successful if the tip of the probe is positioned at a distance less than 5 mm in both axes from the target model and stay stable in place over 5 minutes of ventilation.

CONTACTS AND LOCATIONS:
Locations (1):
- CHUM, Montreal, Quebec, Canada